CLINICAL TRIAL: NCT06672965
Title: A Single Centre, Double Blind, Placebo-controlled Clinical Study Design in Healthy Subjects to Evaluate the Efficacy of Dietary Supplement to Alleviate Stress in Subjects with Mild to Moderate Stress
Brief Title: A Clinical Study to Evaluate the Efficacy of Dietary Supplement to Alleviate Stress Versus Placebo in Subjects with Mild to Moderate Levels of Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RIGCLI22M
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-09

CONDITIONS: Evaluations, Diagnostic Self

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo was prepared as a capsule composed of excipients only (stearic acid and natural caramel color to match the mg weight of the combination supplement capsule). Take two (2) capsules daily with water.
  Interventions: Dietary Supplement: Placebo
- Calming supplement (Active Comparator): The combination supplement was prepared to deliver 600 mg of Lemon Balm extract, 100 mg of Magnolia Bark extract (containing 40 mg of honokiol) and 200 mg L-theanine daily in 2 capsules with water.
  Interventions: Dietary Supplement: anti-stress supplement

INTERVENTIONS:
Dietary Supplement: anti-stress supplement — The anti-stress supplement was developed to provide relief from anxiety and depression levels.Subjects were given 60 capsules of calming supplement (30-day supply) and instructed to take two capsules each day orally with water.
  Arms: Calming supplement
Dietary Supplement: Placebo — Subjects were given 60 capsules of placebo (30-day supply) and instructed to take two capsules each day orally with water.
  Arms: Placebo

SUMMARY:
A single centre, double blind, placebo-controlled clinical study design in healthy subjects to evaluate the efficacy of dietary supplement to alleviate stress in subjects with mild to moderate stress

ELIGIBILITY:
Inclusion Criteria:

1. Must complete pre-study assessment questionnaire and have a minimum stress level score of ≥14.
2. The subject is a healthy male or female 25-55 years of age at the time of informed consent.
3. The subject must have a BMI of ≥18.5 and ≤30.0 kg/m2 and be willing to have their height and weight measured.
4. No reported history of psychological or mental disorders.
5. Free of anti-depressants/anti-anxiety/mood enhancing/recreational drugs (e.g., marijuana, THC, CBD) intake for at least 6 months prior to screening.
6. Free of any 'over the counter' or prescribed medications except for female participants taking contraceptive pills.
7. Agree to abstain from smoking, vaping, or using recreation drugs (e.g., marijuana, THC, CBD) during the study.
8. Willing and able to give informed consent.

Exclusion Criteria:

1. Resting systolic blood pressure above 140 mmHg or a diastolic blood pressure above 90 mmHg at baseline visit.
2. Having taken pharmaceutical products within the last 3 months to help to relieve sleep disturbances or physiological stress.
3. Having taken dietary supplements within the last 3 months to help relieve sleep disturbances or physiological stress.
4. Having taken anti-depressants/anti-anxiety/mood enhancing/ recreational drugs (e.g., marijuana) within 6 months prior to screening.
5. Having smoked, vaped, or used recreational drugs (e.g., marijuana, THC, CBD) within the last 6 months prior to screening.
6. Having any known chronic skin conditions that may be exacerbated with using a topical product.
7. Pregnant, planning to become pregnant or nursing.
8. Any known allergy or intolerance to any of the ingredients contained in supplements or topical product.
9. Individuals with sunburn, moderate to pronounced suntan, uneven skin tones, tattoos, scars or other disfiguration, dilated vessels or other conditions on the test area that might influence the test results.
10. Any disease or condition of the skin that the examining investigator deems inappropriate for participation, including rosacea, eczema, and atopic dermatitis.
11. Individuals currently taking certain medications which in the opinion of the investigators may interfere with the Study. This would include but not be limited to routine high dosage use of anti-inflammatory drugs (aspirin, ibuprofen, corticosteroids) immunosuppressive drugs or antihistamine medications (steroid nose drops and/or eye drops are permitted), and insulin, antihypertensive drugs, antibiotics, or other topical drugs at the test sites.
12. Individuals who have routinely used an alpha-hydroxy-acid (AHA) or a betahydroxy-acid (BHA) containing product within two weeks or Retin-A®, Retin-A Micro®, Renovar®, Differin®, Avita®, Tazorac®, or Soriatane® within one month of the Study start or have taken Accutane® within one year of the Study start.
13. Individuals who have used Retinol in the last six months.
14. Individuals with inflammatory acne lesions (i.e., papules, pustules, cysts, nodules) at the test site.
15. Individuals with known allergies to skin treatment products or cosmetics, toiletries, and/or topical.
16. Individuals taking high dose biotin (i.e., >5 mg / > 5000 μg per day).
17. Individuals who work night shifts.

Ages: 40 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Assessment of anxiety using Hamilton Anxiety Rating Scale (HAM-A) scale | 30 days
  Hamilton Anxiety Rating Scale (HAM-A) (1) was assessed using a questionnaire and scored on a scale of 0 to 4, with 0 (no presence of anxiety) to 4 (severe anxiety). (1) Hamilton, M. The assessment of anxiety states by rating. Br. J. Med. Psychol. 1959, 32, 50-55.
Assessment of depression using Hamilton Depression Rating Scale (HDRS) scale | 30 days
  Hamilton Depression Rating Scale (HDRS) (1) was assessed using a questionnaire and scored using a scale of 0 to 20, with 0-7 (within normal range or remission) while a score of 20 (indicating moderate depression.
  (1) Hamilton, M. A rating scale of depression. J. Neurol. Neurosurg. Psychiatry, 1960, 23, 56-62.
Assessment of perception of stress in subjects that experience moderate levels of stress using Perceived Stress Scale (PSS) | 30 days
  Perceived stress was assessed with Perceived Stress Scale (PSS) using a validated questionnaire on a score of 0 to 40, with 0 (no stress) and 20 or above (higher perceived stress) at day 1, day 7 and at day 30.

SECONDARY OUTCOMES:
Assessment of mood using Profile of Mood States (POMS) scale | 30 days
  Assessment of Profile of Mood States (POMS) was measured on a 5 point scale of 0 to 5, with 0 (not at all moody) to 4 (extremely moody),
Assessment of sleep using Restorative Sleep Questionnaire, Weekly (RSQ-W) version scale | 30 days
  Restorative Sleep Questionnaire, Weekly (RSQ-W) is a nine-item survey that measures how restful a person feels after sleeping for the past week. The RSQ-W scale scores range from 0-100, with higher scores indicating more restorative sleep. To convert the average score to a 0-100 scale, use the formula: RSQ-W Total Score = {RSQ-W Average Score Across Completed Items - 1.0}*25.

CONTACTS AND LOCATIONS:
Locations (1):
- PCR Corp, Manchester, United Kingdom